CLINICAL TRIAL: NCT03359655
Title: A Randomised Trial for Postoperative Pain After Rectal Misoprostol or Rectal Hyoscine Administration
Brief Title: A Trial for Peroperative Procedure and Postoperative Pain After Rectal Misoprostol or Rectal Hyoscine Administration
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bezmialem Vakif University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Diagnostic
Other Study IDs: 2017-6-
Record Dates: First submitted 2017-11-07; First posted 2017-12-02 (Actual); Last update posted 2018-12-27 (Actual); Status verified 2018-12

CONDITIONS: Hysteroscopic Surgery; Pain, Postoperative
Keywords: misoprostol; hyoscine butyl bromide; cervical dilatation; cervical ripening; hysteroscopy; pain
MeSH Terms: conditions — Pain, Postoperative; Pain | interventions — Misoprostol; Butylscopolammonium Bromide

STUDY DESIGN:
Intervention Model Description: Three group parallel design
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Double blind masking
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Rectal misoprostol (Active Comparator): 200 mcg of misoprostol will be administered rectally- 2 hours previously. This intervention will be performed by a third party health professional who will be blinded to the procedure.
  Interventions: Drug: Misoprostol
- Rectal hyoscine butyl bromide (Active Comparator): 10 mg hyoscine butyl bromide administered rectally- 2 hours previously. This intervention will be performed by a third party health professional who will be blinded to the procedure.
  Interventions: Drug: Hyoscine butyl bromide
- Sham administration (No Intervention): A rectal examination will be performed by a third party health professional who will be blinded to the procedure. No drug will be administered

INTERVENTIONS:
Drug: Misoprostol — Rectal administration 2 jours before the procedure
  Other Names: Cytotec
  Arms: Rectal misoprostol
Drug: Hyoscine butyl bromide — Rectal administration 2 jours before the procedure
  Other Names: Buscopan
  Arms: Rectal hyoscine butyl bromide

SUMMARY:
Dilatation of the cervix is necessary before operative hysteroscopic procedures. This dilatation with Hegar dilators has certain difficulties and is associated with pain. Cervical priming with various substances soften the cervix, ease the entry for the operation and decrease complications such as uterine perforation.

The investigators aimed to compare rectally administered "misoprostol" and" hyoscine butyl bromide" with sham protocol.

DETAILED DESCRIPTION:
The study is planned as a double blind randomised controlled one centre study. It will take part at a operative gynaecological department of a university hospital. Women who apply to the university clinic who have a medical indication for hysteroscopic surgery will be recruited after informed consent.

Patients included in the study will be allocated to three groups. The intervention arms will be two arms and one sham group. The randomisation will be performed to three groups by a third party who is not involved in the surgical procedures.

Upon initial evaluation, a form evaluating age and other sociodemographic characteristics will be filled out before the scheduled hysteroscopy procedure. After completion of the initial form, rectal tablets will be administered according to the allocated group; two hours previously to the procedure. Hysteroscopy will be under general anaesthesia with a 10 mm hysteroscope during the follicular phase of the menstrual cycle.

During the procedure the duration of the cervical entry and total duration of the operation will be noted. Additionally basal dilatation will be noted.

Two hours after the procedure pain will be documented according to the Visual Analogue Scale which is a ten point scale. A value of "1" indicates "no pain". A value of "10" indicates "excruciating" pain.

ELIGIBILITY:
Inclusion Criteria:

* Reproductive aged women
* Women who are scheduled for hysteroscopy for indications of endometrial polyp, submucous myoma or synaechiae

Exclusion Criteria:

* Women who have undergone hysteroscopy previously
* women who are in menopause

Ages: 18 Years to 55 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Hysteroscopy is an endoscopic surgery for the uterus
Enrollment: 120 (Actual)
Dates: Start 2018-06-11 (Actual); Primary Completion 2018-12-04 (Actual); Study Completion 2018-12-13 (Actual)

PRIMARY OUTCOMES:
Postoperative pain | Postoperative 2 hours
  Two hours after the procedure "postoperative pain" will be documented according to the Visual Analogue Scale which is a ten point scale. A value of "1" indicates "no pain". A value of "10" indicates "excruciating" pain.

SECONDARY OUTCOMES:
Analgesic administration | Postoperative 2 hours
  Need for analgesic administration
Duration of procedure | During the surgery
  Duration of cervical dilatation and total surgery
Ease of cervical dilatation | During the surgery
  Ease of cervical dilatation will be evaluated using a 5 point likert scale.
  1. Very difficult
  2. Difficult
  3. Normal
  4. Easy
  5. Very easy
Initial cervical dilatation | During the surgery
  Initial cervical dilatation will be evaluated using the Hegar dilatator number

CONTACTS AND LOCATIONS:
Overall Officials: Serdar G Aydin, Principal Investigator — Bezmialem Üniversitesi Tıp Fakültesi Hastanesi
Locations (1):
- Bezmialem Vakif University, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
The results will be published
Supporting Information: Study Protocol, CSR
Time Frame: After the study is completed
Access Criteria: The results will be published in a science citation indexed journal